CLINICAL TRIAL: NCT05768373
Title: Clinical Evaluation of Clinpro™ 2.1% Sodium Fluoride Aqueous Solution in the Treatment of Dentin Hypersensitivity
Brief Title: A Comparison Study of Hypersensitivity Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EM-11-050084
Record Dates: First submitted 2023-03-01; First posted 2023-03-14 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Only subject will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 3M™ Clinpro™ Fluoride Aqueous Solution (Experimental): Investigational product.
  Interventions: Device: 3M™ Clinpro™ Fluoride Aqueous Solution
- 3M™ Vanish™ (Active Comparator): Commercialized product
  Interventions: Device: 3M™ Vanish™

INTERVENTIONS:
Device: 3M™ Clinpro™ Fluoride Aqueous Solution — Hypersensitivity treatment. Apply once after baseline measurement of dentin sensitivity.
  Arms: 3M™ Clinpro™ Fluoride Aqueous Solution
Device: 3M™ Vanish™ — Hypersensitivity treatment. Apply once after baseline measurement of dentin sensitivity.
  Arms: 3M™ Vanish™

SUMMARY:
The goal of this clinical trial is to evaluate the effect of 3M™ Clinpro™ Fluoride Aqueous Solution (experimental) on Dentin Hypersensitivity (DHS) in comparison to 3M™ Vanish™ (commercialized, control] in patients who have DHS.

Participants will be asked to complete the following activities:

Undergo a pre-treatment washout period for 3- to 6-weeks (± 4 days) post-enrollment. During this time, the Subject is to only use the provided oral hygiene products.

Hypersensitivity will be assessed prior to (baseline) and immediately after sample application.

Subject will be asked to come to the facility for hypersensitivity assessments at 24 hours, 7 days, and 30 days after the treatment visit.

Researchers will compare 3M™ Clinpro™ Fluoride Aqueous Solution to 3M™ Vanish™ to evaluate if the effect of Clinpro™ on DHS treatment is non-inferior to Vanish™.

DETAILED DESCRIPTION:
After Informed Consent has been obtained, the subjects will be given study supplied oral hygiene products (e.g., toothbrush and toothpaste) to be used immediately after the consent visit and throughout the entire duration of the study.

Subjects will have a minimum wash-out period of 3 weeks followed by 1 treatment visit. At the treatment visit, a pain assessment will be performed (ie, a baseline pain score) in response to both an air-blast stimulus and tactile stimulus. After each stimulus, the Subject should score their pain using a Visual Analog Scale (VAS).

After recording baseline pain scores, Clinpro™ (Treatment arm) or Vanish™ (Control arm) will be applied according to the manufacturer's IFU. Pain in response to air blast and probe test will be assessed using VAS immediately after application of fluoride treatment (within 15 minutes). Pain response will be assessed again at 24 h, 7 d, 21 d and 30 d post-application of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has at least one affected hypersensitive tooth upon air blast stimuli in the cervical area, and baseline pain score of 40 mm and above as assessed by the 100 mm VAS.
2. Subject is at least 18 years old and have a minimum of 20 natural teeth.
3. Subject is willing to withhold desensitizing treatment, including prescription, in-office or over the counter (OTC) desensitizing products, throughout the study period AND withhold during the washout period.
4. Subject agrees to only use the provided toothpaste, toothbrush, and follows all oral hygiene instructions throughout the study period AND follows all oral hygiene instructions during the washout period.
5. Subject is able to understand and willing to sign the Informed Consent, and is willing to return to the study facility for scheduled study visits and recalls.

Exclusion Criteria:

1. Subject has medical (including psychiatric) and pharmacotherapeutic histories that may compromise the protocol - including the chronic use of anti-inflammatory, analgesic (pain), and mind-altering drugs; or analgesic (pain) medications within 48 hours prior to application of treatment.
2. Subject is pregnant (self-reported) or breast feeding.
3. Subject has allergies to product ingredients, eg, rosin, mint flavoring.
4. Subject has systemic conditions that are etiologic or predisposing to dentin hypersensitivity (eg, chronic acid regurgitation).
5. Subject has excessive dietary or environmental exposure to acids at time of screening.
6. Subject had periodontal treatment, bleaching treatments, or orthodontic treatments within previous 3 months or plans to have any other dental treatments during the study period.
7. Subject is enrolled in another clinical trial at the time of screening that would interfere with this study.
8. Subject is, in the opinion of the investigator, unsuitable for enrollment in the study for reasons other than those specified in the above exclusion criteria.

   Individual teeth may not be included that meet any of the following criteria:
9. Study tooth has periodontal probing depth of ≥ 4 mm.
10. Study tooth or the surrounding supporting tissue has any other painful pathology or defects.
11. Study tooth has been restored in the preceding 3 months.
12. Study tooth is an abutment for fixed or removable prostheses or suffers traumatic malocclusion.
13. Study tooth is crowned or extensively restored and the restorations extending into the test area.
14. The tooth has dentin hypersensitivity due to cracked enamel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, Principal Investigator — Loma Linda University, School of Dentistry
Locations (1):
- LOMA LINDA UNIVERSITY, School of Dentistry, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3M™ Clinpro™ Fluoride Aqueous Solution | 3M™ Vanish™
Started | 51 | 50
Completed | 51 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3M™ Clinpro™ Fluoride Aqueous Solution | 3M™ Vanish™ | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.38) | 44.6 (14.00) | 44.2 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 65
  Male | 15 | 21 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 3 | 1 | 4
  White | 34 | 34 | 68
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 101
Air Blast VAS (Visual Analog Scale) baseline [Mean (Standard Deviation); unit: units on a scale] — The baseline pain score upon air blast stimulus was measured using Visual Analog scale (VAS) prior to the sample application.
  The VAS ranges from 0 mm to 100 mm. 0 mm is no pain, and 100 mm is worst pain. Higher scores mean a worse outcome.
  units on a scale | 62.9 (13.33) | 59.8 (9.95) | 61.3 (11.82)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain From Baseline Immediately After Application of Test Product.
Description: Change in sensitivity as assessed using a Visual Analog Scale (VAS, 0 - 100 mm) immediately after exposure to air stimulus relative to baseline.
  The VAS consists of a 100mm line, with two extremes being 0 mm (no pain) and 100 mm (worst pain). Higher scores mean a worse outcome.
Time Frame: Base line and immediately after application (within 15 minutes post-treatment).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3M™ Clinpro™ Fluoride Aqueous Solution | 3M™ Vanish™
Number analyzed (Participants) | 51 | 50
units on a scale | 8.9 (10.26) | 8.6 (8.41)
Statistical Analysis 1: Comparison: 3M™ Clinpro™ Fluoride Aqueous Solution vs 3M™ Vanish™; Test type: Non-Inferiority — This study used a non-inferiority margin of 15 mm; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-3.4 to 4.0] — The difference is 3M Clinpro minus 3M Vanish

2. Primary Outcome: Change in Pain From Baseline 24 Hours Post Application of Test Product.
Description: This is a co-primary endpoint
  Change in sensitivity as assessed using 100-mm Visual Analog Score (VAS) 24 hours after exposure to air stimulus relative to baseline.
  The VAS consists of a 100mm line, with two extremes being 0 mm (no pain) and 100 mm (worst pain). Higher scores mean a worse outcome.
Time Frame: Baseline and 24 hours post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3M™ Clinpro™ Fluoride Aqueous Solution | 3M™ Vanish™
Number analyzed (Participants) | 51 | 50
units on a scale | 12.8 (10.57) | 11.5 (9.43)
Statistical Analysis 1: Comparison: 3M™ Clinpro™ Fluoride Aqueous Solution vs 3M™ Vanish™; Test type: Non-Inferiority — This study used a non-inferiority margin of 15 mm; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-2.6 to 5.3] — The difference is 3M Clinpro minus 3M Vanish

3. Secondary Outcome: Change in Pain From Baseline 7 Days Post Application of Test Product.
Description: Change in sensitivity as assessed using 100-mm Visual Analog Score (VAS) 7 days after exposure to air stimulus relative to baseline.
  The VAS consists of a 100mm line, with two extremes being 0 mm (no pain) and 100 mm (worst pain). Higher scores mean a worse outcome.
Time Frame: Baseline and 7 days post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3M™ Clinpro™ Fluoride Aqueous Solution | 3M™ Vanish™
Number analyzed (Participants) | 51 | 50
units on a scale | 14.6 (13.45) | 12.9 (11.45)
Statistical Analysis 1: Comparison: 3M™ Clinpro™ Fluoride Aqueous Solution vs 3M™ Vanish™; Test type: Non-Inferiority — This study used a non-inferiority margin of 15 mm; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-3.2 to 6.7] — The difference is 3M Clinpro minus 3M Vanish

4. Secondary Outcome: Change in Pain From Baseline 21 Days Post Application of Test Product.
Description: Change in sensitivity as assessed using 100-mm Visual Analog Score (VAS) 21 days after exposure to air stimulus relative to baseline.
  The VAS consists of a 100mm line, with two extremes being 0 mm (no pain) and 100 mm (worst pain). Higher scores mean a worse outcome.
Time Frame: Baseline and 21 days post-treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 3M™ Clinpro™ Fluoride Aqueous Solution | 3M™ Vanish™
Number analyzed (Participants) | 51 | 50
units on a scale | 18.6 (13.69) | 16.4 (12.47)
Statistical Analysis 1: Comparison: 3M™ Clinpro™ Fluoride Aqueous Solution vs 3M™ Vanish™; Test type: Non-Inferiority — This study used a non-inferiority margin of 15 mm; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-3.0 to 7.4] — The difference is 3M Clinpro minus 3M Vanish

5. Secondary Outcome: Change in Pain From Baseline 30 Days Post Application of Test Product.
Description: Change in sensitivity as assessed using 100-mm Visual Analog Score (VAS) 30 days after exposure to air stimulus relative to baseline.
  The VAS consists of a 100mm line, with two extremes being 0 mm (no pain) and 100 mm (worst pain). Higher scores mean a worse outcome.
Time Frame: Baseline and 30 days post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 3M™ Clinpro™ Fluoride Aqueous Solution | 3M™ Vanish™
Number analyzed (Participants) | 51 | 50
units on a scale | 22.1 (16.81) | 20.3 (15.05)
Statistical Analysis 1: Comparison: 3M™ Clinpro™ Fluoride Aqueous Solution vs 3M™ Vanish™; Test type: Non-Inferiority — This study used a non-inferiority margin of 15 mm; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-4.4 to 8.2] — The difference is 3M Clinpro minus 3M Vanish

ADVERSE EVENTS:
Time Frame: AEs will be collected from the time of initial application of control or investigational treatment until end of study visit (30 days post-application).
Description: No adverse event was reported in this study.
Arm/Group | 3M™ Clinpro™ Fluoride Aqueous Solution | 3M™ Vanish™
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 0/51 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT05768373/Prot_SAP_000.pdf